CLINICAL TRIAL: NCT04407143
Title: Study of Acquired Immunity in Patients With Lung Cancer and COVID-19 Infection
Brief Title: Study of the Immunity of Patients With Lung Cancer and COVID-19 Infection
Acronym: SOLID
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 20/04_SOLID
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer; COVID; Corona Virus Infection
Keywords: IgG; coronavirus; COVID-19; lung cancer
MeSH Terms: conditions — Lung Neoplasms; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung cancer+COVID-19: Lung cancer patients infected by COVID-19
  Interventions: Diagnostic Test: IgG test

INTERVENTIONS:
Diagnostic Test: IgG test — IgG+ blood test by ELISA method.

SUMMARY:
Observational, retrospective data collection and prospective IgG analysis, and multicenter study.

The main objective of the study is th description of the characteristics and evolution of patients with lung cancer who have acquired COVID-19 infection.

For the identification of patients who contract COVID-19 infection, the IgG+ blood test by ELISA method will be used.

DETAILED DESCRIPTION:
Non-post-authorization study, retrospective of data collection and prospective of IgG analysis, observational and multicenter.

The study will be extended to all the sites of the Spanish Lung Cancer Group, more than 170 centers and 500 professionals, and it is expected that around 1,500 IgG tests will be carried out.

The study has three phases:

The scope of phase I is the identification of acquired immunity (IgG) in patients with lung cancer, whether or not they have presented symptoms of having suffered from COVID19. In addition, the description of the characteristics and evolution of patients with lung cancer who have contracted COVID-19 infection will be carried out.

For the identification of patients who contract COVID-19 infection, the IgG+ test in blood will be used by ELISA method.

The scope of phase II is the confirmation of the presence of antibodies (IgG) in patients who tested positive in Phase I of the study a few weeks after the first diagnosis made through the SOLID study.

The scope of phase III is the confirmation of the presence of antibodies (IgG) in patients with lung cancer who have been vaccinated with any of the available and authorized vaccines for SARS-COV2 and 6 months after said administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with lung cancer at any stage of the disease
2. Age ≥ 18
3. Patients who have signed the informed consent for this study

Exclusion Criteria:

1. Patients who have not signed or do not wish to sign the informed consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have not signed or do not wish to sign the informed consent for this study
Sampling Method: Non-Probability Sample
Enrollment: 1980 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Description of the characteristics of patients | From the diagnosis of the COVID until the determination of the blood IgGs, up to 10 weeks
  Description of the characteristics and evolution of patients with lung cancer who have contracted COVID-19 infection.

SECONDARY OUTCOMES:
Detection of antibodies (IgG) at 6 months after SARS-COV2 vaccines | From the date of complete SARS-COV2 vaccination administration until 6 month
  Confirmation of the presence of antibodies (IgG) in patients with lung cancer who have been vaccinated with any of the available and authorized vaccines for SARS-COV2 and 6 months after such administration.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Principal Investigator — Hospital Puerta de Hierro de Majadahonda de Madrid
Locations (68):
- Spain (68):
  - Complejo Hospitalario de A Coruña, A Coruña, A Coruña
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Burgos, Burgos, Burgos
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Dr. Josep Trueta, Girona, Girona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario de Jaén, Jaén, Jaén
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Clínica Universidad de Navarra, Madrid, Madrid
  - Hospital de Sanchinarro, Madrid, Madrid
  - Hospital Severo Ochoa, Madrid, Madrid
  - Hospital Universitario Infanta Cristina, Madrid, Madrid
  - Hospital Universitario de Torrejón, Torrejón, Madrid
  - Hospital Universitario Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital General Universitario de Málaga, Málaga, Málaga
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitari i Politécnic La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital La Esperanza, A Coruña
  - Hospital Universitario de Ferrol, A Coruña
  - Hospital Virgen de los Lirios, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Cruces, Bilbao
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital General La Mancha Centro, Ciudad Real
  - Hospital Universitario de Vinalopó, Elche
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Asistencial Universitario de León, León
  - Hospital universitari Arnau de Vilanova, Lleida
  - Hospital San Pedro, Logroño
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Móstoles, Madrid
  - Hospital Universitario del Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital Costa del Sol, Málaga
  - Complejo Hospitalario Universitario de Ourense Santa María Nai, Ourense
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Clínica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Sant Joan de Reus, Reus
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - Hospital Sant Pau i Santa Tecla, Tarragona
  - Hospital Arnau de Vilanova, Valencia
  - Hospital de Manises, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Lluís Alcanyís, Valencia
  - Hospital Universitario Río Ortega, Valladolid
  - Complejo Hospitalario Zamora, Zamora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Provencio M, Estival A, Franco F, Lopez-Vivanco G, Saigi M, Arasanz H, Diz P, Carcereny E, Garcia J, Aguado C, Mosquera J, Iruarrizaga E, Majem M, Bosch-Barrera J, Mielgo-Rubio X, Guirado M, Juan-Vidal O, Blasco A, Lucia Gozalvez C, Del Barrio A, De Portugal T, Lopez-Martin A, Serrano G, Campos B, Rubio J, Catot S, Esteban B, Marti-Ciriquian JL, Del Barco E, Calvo V; Spanish Lung Cancer Group (SLGC/GECP). Immunogenicity of COVID-19 vaccines in lung cancer patients. Lung Cancer. 2023 Oct;184:107323. doi: 10.1016/j.lungcan.2023.107323. Epub 2023 Aug 9. PMID 37639820
- [Derived] Provencio M, Rodriguez-Abreu D, Ortega AL, Serrano G, Aguado C, Franco F, Gutierrez V, Lopez Vivanco G, Guirado M, Benitez G, Estival A, Calvo V, Jimenez B, Arasanz H, Coves J, Majem M, Massuti B, Vazquez S, Juan-Vidal O, Collazo-Lorduy A, Gozalvez CL, Del Barco E, Rosero A, Bosch-Barrerra J, Moreno MA, Mielgo-Rubio X, Villa JC, Lopez-Martin A, Cordoba JF, de Asis Aparisi F, Zafra M, Mosquera J, Perez Altozano J, Nadal E, Catot S, Balsalobre J, de Portugal T, Martin P, Cuesta de Juan S, Cobo M. Seroprevalence and immunological memory against SARS-CoV-2 in lung cancer patients: the SOLID study. Transl Lung Cancer Res. 2022 Jan;11(1):53-63. doi: 10.21037/tlcr-21-504. PMID 35242627
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org